CLINICAL TRIAL: NCT05593900
Title: Nurse-to-Family Telehealth for Pediatric Transfers: A Randomized Controlled Pilot Trial
Brief Title: Nurse-To-Family Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1062184
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents have the option to use telehealth to virtually connect with the nurse before transfer
  Interventions: Behavioral: Nurse-to-Family Video Chat
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Nurse-to-Family Video Chat — A Nurse-To-Family Video Chat will be offered to parents/guardians to virtually connect with their post-transfer nurse; this intervention is changing the behavior of how providers deliver healthcare and how parents/guardians engage in their child's care.
  Arms: Intervention

SUMMARY:
This study will be a pilot test of using telehealth to allow nurses to connect with parents/guardians of pediatric patients who are being transferred between hospitals.

ELIGIBILITY:
Inclusion Criteria:

Children who:

* are aged 8 days to <=18 years
* present to a participating community hospital ED
* are accepted for inter-facility transfer to UC Davis
* are assigned to UC Davis unit D10, D7, or T6
* have an English-speaking adult parent/guardian at the bedside

Exclusion Criteria:

* does not have an English-speaking adult parent/guardian at the bedside

For parent surveys --

Inclusion Criteria:

* are parents/guardians of the eligible patients (described above)
* are age 18 years and older
* are English-speaking

Exclusion Criteria:

* are age less than 18 years
* have a preferred language that is other than English

Min Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Rosenthal JL, Hoyt-Austin AE, Ketchersid A, Sanders A, Harper TA, Tancredi DJ, Young HM, Romano PS, Marcin JP. Nurse-to-family telehealth for pediatric transfers: protocol for a feasibility and pilot cluster randomized controlled trial. Pilot Feasibility Stud. 2023 Apr 11;9(1):57. doi: 10.1186/s40814-023-01292-4. PMID 37041600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The unit of randomization was the community emergency department (ED). Rationale for randomizing at the ED level was that it decreased contamination in comparison to randomization at the patient level. We used constrained randomization to better balance the intervention and control arms with respect to ED-to-children's hospital distance and pediatric transfer volume. Participants were grouped as families, with one child participant and one parent participant per family.
Units Other Than Participants: community emergency department
Groups:
- Intervention: Among the families who presented to one of the three emergency departments randomized to the intervention arm, parents had the option to use telehealth to virtually connect with the nurse before transfer ("Nurse-to-Family Video Chat"). Thus the intervention was having the option to use the telehealth innovation in addition to usual care. The decision to use telehealth in this trial was encouraged in the intervention arm but remained optional; no nurse or parent was required to use telehealth.
  Nurse-to-Family Video Chat: A Nurse-To-Family Video Chat was offered to parents/guardians to virtually connect with their post-transfer nurse; this intervention was changing the behavior of how providers deliver healthcare and how parents/guardians engage in their child's care.
- Control: Among the families who present to one of the three emergency departments randomized to the control arm, they will receive standard of care (which is not having the option to use the Nurse-to-Family intervention).
Period: Overall Study
Arm/Group | Intervention | Control
Started (77 intervention parents + 77 intervention children = 154 total intervention participants; 39 control parents + 39 control children = 78 total control participants) | 154; 3 community emergency department | 78; 3 community emergency department
Parents | 77; 3 community emergency department | 39; 3 community emergency department
Children | 77; 3 community emergency department | 39; 3 community emergency department
Completed | 154; 3 community emergency department | 78; 3 community emergency department
Not Completed | 0; 0 community emergency department | 0; 0 community emergency department

BASELINE CHARACTERISTICS:
Population: Overall # of baseline participants is 77 intervention families & 39 control families. Each family consisted of 2 participants: a pediatric patient (child) and their parent/guardian. Thus, total # of participants was 154 intervention & 78 control.
  Baseline data includes data of (a) enrolled pediatric patients plus (b) the parent. Data collection used electronic health record (for pediatric patient data) and parent surveys (for parent data). Parent baseline data unknown if survey not completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 77 | 39 | 116
Age, Continuous [Mean (Standard Deviation); unit: years]
  Children | 5.6 (5.4) | 5.2 (5.7) | 5.4 (5.5)
  Parents | 34.7 (9.0) | 34.7 (8.0) | 34.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 19 participants had unknown sex
  Participants
    Children: Female | 26 | 21 | 47
    Children: Male | 51 | 18 | 69
    Parents: number analyzed (Participants) | 63 | 34 | 97
    Parents: Female | 54 | 24 | 78
    Parents: Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall Number of Baseline Participants is presented separately by Children and by Parents.
  Participants
    Children: Hispanic or Latino | 6 | 11 | 17
    Children: Not Hispanic or Latino | 57 | 15 | 72
    Children: Unknown or Not Reported | 14 | 13 | 27
    Parents: Hispanic or Latino | 14 | 13 | 27
    Parents: Not Hispanic or Latino | 48 | 20 | 68
    Parents: Unknown or Not Reported | 15 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall Number of Baseline Participants is presented separately by Children and by Parents.
  Participants
    Children: American Indian or Alaska Native | 0 | 0 | 0
    Children: Asian | 1 | 0 | 1
    Children: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Children: Black or African American | 3 | 2 | 5
    Children: White | 19 | 3 | 22
    Children: More than one race | 2 | 0 | 2
    Children: Unknown or Not Reported | 51 | 34 | 85
    Parents: American Indian or Alaska Native | 3 | 0 | 3
    Parents: Asian | 3 | 7 | 10
    Parents: Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
    Parents: Black or African American | 5 | 6 | 11
    Parents: White | 36 | 9 | 45
    Parents: More than one race | 7 | 2 | 9
    Parents: Unknown or Not Reported | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Assignment Adherence
Description: Percentage of eligible patients for whom the protocol assignment (telehealth vs standard of care) was followed
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 154 | 78
Participants | 4 | 76

2. Secondary Outcome: Fidelity: Percentage of Telehealth Initiated Before Arrival
Description: Whether or not a telehealth connection was initiated prior to patient's arrival to UC Davis hospital. Time of telehealth initiation, if applicable, was obtained from the ExtendedCare (telehealth platform) reporting system. Time of patient arrival was obtained from the electronic health record.
Time Frame: Day 0
Population: Telehealth connection was initiated among 4 intervention arm participants. This measure was not applicable for the Control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 0
Participants | 4 |

3. Secondary Outcome: Survey Completion Rate (%)
Description: Percentage of completed surveys among eligible respondents
Time Frame: Day 0
Population: Surveys sent to one parent/guardian per family.
Measure: Mean (95% Confidence Interval); unit: percentage of completed surveys
Arm/Group | Intervention | Control
Number analyzed (Participants) | 77 | 39
percentage of completed surveys | 81.8 [71.4 to 89.7] | 87.2 [72.6 to 95.7]

4. Other Pre Specified Outcome: Family-Centered Care
Description: Unit of measure: mean score Measure/Tool: Family-Centered Care Experience (FACCE)
Time Frame: Day 0
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Family Experience
Description: Unit of measure: mean score Measure/Tool: Emergency Department CAHPS (Consumer Assessment of Healthcare Providers and Systems) 2 items measuring overall experience
Time Frame: Day 0
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Parent Acute Stress
Description: Unit of measure: mean score Measure/Tool: (parent-reported survey) PROMIS 7-item Emotional Distress: Anxiety
Time Frame: Day 0
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Parent Distress
Description: Unit of measure: mean score Measure/Tool: (parent-reported survey) PROMIS 7-item Emotional Distress: Anxiety
Time Frame: Day 30
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Level of Care
Description: Unit of measure: Percentage of subjects with change in level of care among eligible subjects.
  subjects
  - Definition: (chart review dichotomous outcome) Switching from an acute care unit or service to an intensive care unit or service, and vice versa.
Time Frame: Day 0
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Minimal risk intervention.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/39
Other Adverse Events (participants affected / at risk) | 0/77 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT05593900/Prot_SAP_000.pdf